CLINICAL TRIAL: NCT04339322
Title: Characteristics and Outcome of COVID-19 Among Egyptian Patients
Brief Title: Characteristics and Outcome of Coronavirus Disease 2019 (COVID-19) in Egypt
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidi Karam, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: COVID-19 in Egypt
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Characteristics Diseases; Outcome, Fatal
Keywords: Covid-19; characteristics; Outcome; Egypt
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Covid-19: Patients with clinical presentation and confirmed as Covid-19 according to the definition of Egyptian Ministry of Health
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Follow up to assess the outcome until complications, improvement, death or being transferred to another quarantine hospital.

SUMMARY:
The World Health Organization (WHO) has recently declared coronavirus disease 2019 (Covid-19) a public health emergency of international concern. Egypt is one of the countries that has been infected by Covid-19. The characteristics of clinical presentation, laboratory and radiological data are not yet studied. Outcomes of covid-19 in Egypt also have not been described yet.

DETAILED DESCRIPTION:
Patients admitted to Assiut University hospital, Al Rajhi liver hospital and other covid-19 Quarantine hospitals will be included. The characteristics of patients will be described such as demographic data; age, sex,history of contact to COVID-19 patients or traveling abroad and their clinical manifestation such as fever,cough,shortness of breath, sore throat, diarrhea. Laboratory data will also be included such as blood picture,D-Dimer, serum ferritin, creatinine, liver enzymes, oxygen saturation and covid-19 polymerase chain reaction (PCR). Radiological data will be described as regarding chest X-ray and/or computed tomography.

Patients will be followed until complications, improvement, transfer to another hospital or death and their outcome will be described.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Covid-19 .

Exclusion Criteria:

* Patients refuse to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical presentation and confirmed as Covid-19 according to the definition of Egyptian Ministry of Health.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Demographics of Coronavirus Disease 2019 (COVID-19) in the cohort group | 2 months
  Sheet recording age, sex, co-morbidity,history of contact
Clinical manifestations of Coronavirus Disease 2019 (COVID-19) | 2 month
  Sheet recording symptoms and signs
Laboratory data of included Coronavirus Disease 2019 (COVID-19) cohort | 2 months
  blood picture,D-Dimer, creatinine, liver enzymes
Radiological features of Coronavirus Disease 2019 (COVID-19) cohort | 2 month
  Chest x-ray and/or Computed tomography

SECONDARY OUTCOMES:
outcomes of Coronavirus Disease 2019 (COVID-19) infection in the cohort group | 1 week
  Data recording of the outcomes of treatment

IPD SHARING:
Plan to Share IPD: No
The data prescribed in the study